CLINICAL TRIAL: NCT04486677
Title: Caring Cards to and From Veterans: Feasibility and Acceptability of a Peer Approach to Suicide Prevention and Recovery
Brief Title: Caring Cards to and From Veterans: A Peer Approach to Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3445-P
Record Dates: First submitted 2020-06-29; First posted 2020-07-24 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Feasibility; Acceptability; Thwarted Belongingness; Perceived Burdensomeness; Suicide Risk; Social Connectedness
Keywords: Veterans; Suicide; Thwarted belongingness; Perceived burdensomeness; Social connectedness
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: The current study is a single-site, 2-year pilot trial that employs an open-trial, pre/post research design. This study's primary aim is to establish the feasibility and acceptability of Caring Cards for Veterans, a peer-centered intervention that facilitates suicide prevention and social connectedness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caring Cards Group (Other): Group of Veteran card-makers.
  Interventions: Behavioral: Caring Cards Group
- Caring Cards Recipients (Other): Group of Veteran card-recipients.
  Interventions: Behavioral: Caring Cards Recipients

INTERVENTIONS:
Behavioral: Caring Cards Group — Group of Veteran card-makers.
  Arms: Caring Cards Group
Behavioral: Caring Cards Recipients — Group of Veteran card-recipients.
  Arms: Caring Cards Recipients

SUMMARY:
Veteran suicide is a national problem; social disconnection is an important contributor to suicide risk. This pilot study will recruit Veterans to take part in a peer-centered intervention called Caring Cards (CC). CC gives Veterans who have a history of increased suicide risk the opportunity to make cards that are then sent to Veterans who are currently at high-risk for suicide. This study will directly benefit Veterans and contribute to the quality of services provided by VA by creating a safe, creative space for Veterans with lived experience related to suicide risk to join together to provide messages of hope, community, and resilience to their peers at risk for suicide. Helping Veterans support one another provides a bridge for social connection, which may help prevent Veteran suicide. This intervention may also improve Veterans' satisfaction with VA healthcare and engagement with mental health treatment.

DETAILED DESCRIPTION:
There is a strong need to develop, evaluate, and implement translatable interventions aimed at reducing Veteran suicide. Caring contacts for suicide prevention (i.e., staff send supportive letters to patients following psychiatric inpatient stays) is an empirically supported, low-cost method for meaningfully reducing suicide risk and hospitalization readmissions and, has been studied and applied in Veterans/VA settings. Peer support (i.e., persons with lived mental health experience) in mental health recovery is another empirically supported approach. Peers' involvement in mental healthcare improves patients' social functioning and community integration, as well as reduces self-stigma and functional impairment. This study focuses on the Caring Cards (CC) intervention, which is a novel integration of caring contacts and peers. In CC, outpatient Veterans with lived mental health experience (peers) create hope-filled and inspiring cards that are then sent to other Veterans struggling with mental health concerns. By design, CC increases social connectedness among participants to reduce suicide risk, which is strongly associated with social disconnectedness. Indeed, there are two evidence-based social risk factors of suicide: thwarted belongingness (TB; feeling like one does not belong) and perceived burdensomeness (PB; feeling as though one's existence is a burden on others). CC combines both caring contacts and peers to specifically target reductions in TB and PB by increasing social connectedness. This study aims to establish the feasibility and acceptability of CC. The investigators' initial quality improvement project provided strong preliminary evidence for the feasibility and acceptability of the CC. The current study is a single-site, 2-year pilot trial that employs an open-trial, pre/post research design. The investigators propose to recruit outpatient Veterans with a history of high suicide risk to make up the CC group and serve as the card-makers (CMs). The investigators will recruit outpatient Veterans who are currently at high-risk for suicide to be the card-recipients (CRs). The primary outcome (Aim 1) is to establish feasibility and acceptability of CC. Aim 2 will examine CC's ability to reduce the primary outcomes (TB and PB) among CMs and CRs. Aim 3 will preliminary evaluate CC's ability to increase social connectedness, as well as reduce suicide risk (i.e., suicidal ideation and behavior) among CMs and CRs. CMs will meet in weekly groups, each for six months, over the course of one year; CRs will receive a total of six cards, one per month. Monthly meet-up groups will also be an optional venue for CMs and CRs to meet each other in-person. Baseline and follow-up assessments will be completed at start and one month after final group for CMs, or one month after the final card for CRs. This project builds on the investigators' preliminary data which indicate that Veteran CMs are interested in and find participating in CC groups highly meaningful, and Veteran CRs enjoy receiving the cards, want to receive more, and describe them as inspirational and empowering. This project is innovative in its utilization of peers to facilitate suicide prevention and social recovery among Veterans at risk for suicide by specifically targeting TB and PB. It is also unique in that it simultaneously targets two populations (outpatient Veterans with a history of, and those with current suicide risk), which have not previously been examined with traditional caring contacts. This research directly responds to the National Prioritized Research Agenda for Suicide Prevention. This study directly supports RR&D's mission and is aligned with VA's 2018-2028 National Strategy for Preventing Veteran Suicide. The investigators expect that these data will inform best practices in suicide prevention and social recovery for Veterans at risk for suicide.

ELIGIBILITY:
Inclusion Criteria:

* For card-makers:

  * VA San Diego Healthcare System (VASDHS) Veteran with an inactive high-risk flag,
  * 18 years of age or older,
  * access to transportation to attend the group (if held in person)
  * if groups are held remotely due to COVID-19, access to reliable technology and WiFi to participate via WebEx
  * decisional capacity.
* For card-recipients:

  * VASDHS Veteran with an active high-risk flag,
  * 18 years of age or older, and
  * decisional capacity.

Exclusion Criteria:

-For card-makers and recipients:

* the absence of a mailing address or working phone number,
* inability to read and writer in English, and
* previous or current experience with Caring Cards.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Granholm, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
One or more data sets without personal identifiers will be generated during the data analysis phase of this study. The data sets will include all data underlying any publications generated by this study and therefore these will be sufficient to reproduce or verify any published findings. Data sets without personal identifiers will be generated. Any HIPAA identifiers, or combinations of variables that could be used for re-identification, will be excluded, as will any proprietary information. The plan does not include any access to individually identifiable or proprietary data. Therefore, this plan will ensure the protection of personal privacy, the confidentiality of individually identifiable private information, and the security of proprietary data and information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Final data sets underlying publications resulting from this research will be shared upon written request. Requests for access must be made in writing signed by a requestor from the United States and include an email address for delivery and an assurance that the recipient will not attempt to identify or re-identify any individual. The request should reference the publication underlying the request. Requests may be made to the Principal Investigator/lead point-of-contact for the publication. If the investigator leaves the VASDHS the requests may be sent to the Associate Chief of Staff for Research.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caring Cards Group | Caring Cards Recipients
Started | 30 | 50
Completed | 21 | 34
Not Completed | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caring Cards Group | Caring Cards Recipients | Total
Number analyzed (Participants) | 30 | 50 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 47 | 75
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 20 | 35 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 22 | 29 | 51
  Unknown or Not Reported | 2 | 14 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 11 | 15
  White | 22 | 29 | 51
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 50 | 80
Era of Military Service [Count of Participants; unit: Participants]
  Persian Gulf War | 26 | 45 | 71
  Post-Vietnam | 3 | 2 | 5
  Vietnam | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: Feasibility will be measured by the proportion of Veterans 1) referred for screening, 2) determined eligible, 3) enrolled/completed baseline, and 4) complete follow-up assessments.
Time Frame: Through study completion, approximately 1 year, 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Caring Cards Group | Caring Cards Recipients
Number analyzed (Participants) | 380 | 370
Participants
  referred for screening | 242 | 234
  determined eligible | 212 | 233
  enrolled/completed baseline | 30 | 50
  complete follow-up assessments | 21 | 34

2. Primary Outcome: Intervention Satisfaction Questionnaire (Acceptability)
Description: Intervention Satisfaction Questionnaire will be collected from participants following intervention delivery to measure acceptability of the Caring Cards intervention.
Time Frame: Through study completion, approximately 1 year, 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Caring Cards Group | Caring Cards Recipients
Number analyzed (Participants) | 21 | 34
Participants
  Perception of benefit | 13 | 21
  Recommend to other Veterans | 11 | 22

3. Secondary Outcome: Interpersonal Needs Questionnaire (INQ-15)
Description: At baseline and follow-up, Veterans will complete the INQ-12 to assess for thwarted belongingness and perceived burdensomeness. Each item on the INQ is rated on a 1-7 Likert scale so the full range of the measure is 12-105, with scores meaning higher thwarted belongingness and perceived burdensomeness (i.e., a worse outcome).
Time Frame: Change from baseline, an average of 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caring Cards Group | Caring Cards Recipients
Number analyzed (Participants) | 21 | 34
score on a scale
  Baseline | 39.19 (24.07) | 54.35 (21.15)
  9 month follow up | 36.67 (21.16) | 49.18 (23.13)

4. Secondary Outcome: Suicide Risk
Description: At baseline and follow-up, Veterans' suicide risk was assessed using the Beck Scale for Suicide Ideation (BSSI). It is a 19 item measure on a 0-2 point scale for a range of 0-38, with higher scores indicating higher suicidal ideation or worse outcomes. There are two additional questions about suicide attempts that are not included in the total score.
Time Frame: Change from baseline, an average of 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caring Cards Group | Caring Cards Recipients
Number analyzed (Participants) | 21 | 34
score on a scale
  Baseline | 5.95 (5.83) | 11.50 (6.33)
  9 month follow up | 6.10 (4.55) | 10.21 (7.31)

5. Secondary Outcome: NIH Toolbox Adult Social Relationships Scales
Description: At baseline and follow-up, Veterans will complete the NIH Toolbox Adult Social Relationships Scales to assess social connectedness. There were three subscales included: Perceived Rejection, Loneliness, and Emotional Support. Each includes items rated on a 1-5 scale. Perceived Rejection is 8 items for a range of 8-40, Loneliness is 5 items for a range of 5-25, and Emotional Support is 8 items for a range of 8-40. Higher scores are associated with worse outcomes for Perceived Rejection and Loneliness, while higher scores are associated with better outcomes for Emotional Support.
Time Frame: Change from baseline, an average of 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caring Cards Group | Caring Cards Recipients
Number analyzed (Participants) | 21 | 34
score on a scale
  Baseline (Perceived Rejection) | 17.52 (9.10) | 21.79 (8.29)
  Follow up (Perceived Rejection) | 18.91 (8.58) | 18.41 (8.37)
  Baseline (Loneliness) | 14.19 (6.42) | 18.59 (4.83)
  Follow up (Loneliness) | 13.38 (5.81) | 17.29 (6.59)
  Baseline (Emotional support) | 31.19 (8.69) | 26.18 (8.69)
  Follow up (Emotional support) | 31.52 (9.67) | 29.47 (10.50)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of participant entry into the study until final assessment, which averaged 9 months.
Description: Systematic method:
  Veterans with active high-risk suicide flags are closely monitored and assessed by VA Suicide Prevention Coordinator (SPCs). At baseline and follow-up, participants are administered two suicide screening measures. Veterans who screen positive immediately meet with a licensed provider. Any new suicidal behavior will be documented in a VA-required report. Trained staff will assess and refer Veterans who require immediate medical attention or psychiatric treatment.
Arm/Group | Caring Cards Group | Caring Cards Recipients
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/50
Other Adverse Events (participants affected / at risk) | 0/30 | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caring Cards Group (N=30) | Caring Cards Recipients (N=50)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) — These two attempts resulted in hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caring Cards Group (N=30) | Caring Cards Recipients (N=50)
Suicide attempt (Psychiatric disorders) | 0 (0) | 6 (6) — These attempts did not result in hospitalization; participants remained stable in outpatient treatment with suicide prevention coordinator oversight.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT04486677/Prot_001.pdf
  • Informed Consent Form (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04486677/ICF_000.pdf